CLINICAL TRIAL: NCT01311388
Title: Construction of the "Patient-Centered"Molecular Pathology Diagnostic Center
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Ta Chiu, Taipei Medical University-Center of Excellence For Cancer Research, TMU-CECR
Other Study IDs: 99049
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators want to achieve the goal of diagnosis in early phase, accurate treatment and existence for a long period in order to screen in early phase, diagnose in clinical trial, choose treatment and evaluate prognosis of cancers by establishing molecular pathology tools.

DETAILED DESCRIPTION:
This research is going to discuss the biomarker expression of common malignant neoplasm (tumor)among Taiwanese, such as large intestine rectal cancer, breast cancer, prostate gland cancer, lung cancer, oral cancer, gastric cancer, liver cancer, cervical cancer, cancer of the womb, ovarian cancer, carcinoma of urinary bladder, kidney cancer and so on.

The investigators hope to find the biomarker of common tumors among Taiwanese in order to develop the tools of tumor screening, diagnosis, treatment methods and prediction prognosis

ELIGIBILITY:
Inclusion Criteria:

* above 20 years old
* all kinds of cancer patients

Exclusion Criteria:

* under 20 years old
* none cancer patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-08; Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ta Chiu, Principal Investigator — TMU-CECR
Locations (1):
- TMU-CECR, Taipei, Taiwan